CLINICAL TRIAL: NCT04581460
Title: Primitive Immunodeficiency and Pregnancy
Acronym: PREPI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200747; 2020-A01781-38 (Other: IDRCB number)
Record Dates: First submitted 2020-09-21; First posted 2020-10-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Primary Immune Deficiency
Keywords: Primary immune deficiency; Obstetric experiences; Infectious complications; Pregnancy; Postpartum; Contraception
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients entered in the register of the reference Center for Hereditary Immune Deficits (CEREDIH), hospital Necker-Enfants Malades, Paris, and having reported at least one pregnancy or attempted pregnancy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire intended for patients on the course of pregnancy and postpartum, the neonatal period and contraceptive modalities.

SUMMARY:
The management of patients with primary immune deficiency is increasingly codified, however contraception and pregnancy have not yet extensively studied or codified, and the medical monitoring and the prevention of infectious complications thus remains at the discretion of the practitioner.

The aim the research is to study the obstetric features and outcome of patients with primary immune defects.

DETAILED DESCRIPTION:
Primary immune deficiencies constitute a large group of immune system disorders of genetic origin which can associate, to varying degrees, an increased susceptibility to infections and immunopathological manifestations: allergy, inflammation, autoimmunity, lymphoproliferation, tumors malignant.

Although their prevalence remains underestimated, there has been an increase in the number of cases diagnosed in the past 10 years. The national average prevalence is 8.6 patients per 100,000 inhabitants and the diagnostic incidence is 400 new cases per year in France. Major improvement in the management of primary immunodeficiencies have drastically changed patients outcome. Most patients now reach adulthood and the possibility of carrying out a pregnancy project, that has already reported for patients suffering from hypogammaglobulinemia or variable common immune deficiency, is now increasingly reported for other types of inherited immunodeficiencies. Whereas the management of patients with hereditary immunodeficiencies is increasingly codified, contraception and pregnancy have not yet been the subject of recommendations: medical monitoring and the prevention of infectious complications thus remain at the discretion of the practitioner.

The aim the research is to study the obstetric experiences of patients with a primary immune deficiency, paying particular attention to infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman with Hereditary Immune Deficits and entered in the reference Center for Hereditary Immune Deficits (CEREDIH, hospital Necker-Enfants Malades, Paris) register
* Patient having reported at least one pregnancy or attempted pregnancy
* Patient not opposing to participation in research

Exclusion Criteria:

- Refusal to participate of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients with any inherited immune defect included in the CEREDIH national cohort
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Infectious events | 18 months
  Number of infectious events at any time during pregnancy and post-partum

SECONDARY OUTCOMES:
Infectious gynecological complications | Up to 50 years
  Number of infectious gynecological complications during contraception
Onset of pregnancy | Up to 50 years
  Number of pregnancies during reproductive age period
Pregnancy outcomes | Up to 9 months
  Rate of early or late miscarriage, completed pregnancy, live birth and childbearing
Treatments | 9 months
  Number of treatments aiming at preventing infections
Screening of infections | 9 months
  Presence/absence of screening for infections
Occurrence of obstetric complications | 9 months
  Rate of obstetric complications
Contraception effectiveness | Up to 50 years
  Number of unwanted pregnancies
Contraception complications | Up to 50 years
  Number of non-infectious complications of contraception
Deaths and complications in the neonatal period | 3 months
  Number of complications during neonatal period, including death

CONTACTS AND LOCATIONS:
Overall Officials: Elise Mallart, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Caroline Charlier-Woerther, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Nizar Mahlaoui, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mallart E, Francoise U, Driessen M, Blanche S, Lortholary O, Lefort A, Caseris M, Fischer A, Mahlaoui N, Charlier C; PREPI study group. Pregnancy in primary immunodeficiency diseases: The PREPI study. J Allergy Clin Immunol. 2023 Sep;152(3):760-770. doi: 10.1016/j.jaci.2023.05.006. Epub 2023 May 18. PMID 37210041